CLINICAL TRIAL: NCT00071500
Title: A Novel Technology to Improve HIV Medication Compliance
Brief Title: An Electronic Pillbox for People With HIV
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Vesta Brue, MBA, Medsignals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R43AI052634-01 (NIH); 1R43AI052634-01 (NIH)
Record Dates: First submitted 2003-10-24; First posted 2003-10-28 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: Compliance; Adherence; Computerized; Electronic Pillbox; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Patient Compliance

STUDY DESIGN:
Who Masked: Care Provider

ARMS (3):
- 1 (Experimental): Participants will use MedSignals with all of its features
  Interventions: Device: MedSignals™
- 2 (Experimental): Participants will use MedSignals with only alarm features
  Interventions: Device: MedSignals™
- 3 (No Intervention): Participants will not use any device

INTERVENTIONS:
Device: MedSignals™ — An electronic device that is used to improve medication compliance among HIV patients. It allows convenient storage and transport of antiretroviral medications and functions as an aid to compliance by incorporating reminding alarms at dosing times and usage reporting functions.
  Arms: 1; 2

SUMMARY:
Anti-HIV drug regimens can be very complicated. This study will evaluate a new electronic pillbox designed to help people take their anti-HIV drugs correctly.

DETAILED DESCRIPTION:
Recent advances in antiretroviral therapy have allowed for almost complete inhibition of viral replication in HIV-infected individuals. Unfortunately, the ability of the virus to rapidly mutate and become resistant to treatments necessitates the administration of multiple medications, in complex dosing schedules, to maintain viral suppression. Although adherence to these complicated treatment regimens is paramount, even the most vigilant persons often have difficulty maintaining these protocols for extended periods of time.

MedSignals™ is an electronic device that was designed to improve medication compliance among HIV patients. It allows convenient storage and transport of antiretroviral medications and functions as an aid to compliance by incorporating reminding alarms at dosing times and usage reporting functions. The system alarms at pill times, records pill-taking, communicates usage data to servers, and displays progress charts on personalized web pages. Four separately-controlled compartments are easily set for number of dosings per day and number of pills at each dosing. Thereafter, all alarms are relative to last lid openings, assuring intake is optimally spaced. Additional menu options can be set to advise when lids are opened, such as "take with food." Lid openings are time-stamped in memory. The cradle is permanently plugged into telephone and electrical lines for uploading of data and recharging, but the pillbox is portable and pocket-sized. Every day, sensors detect a phone line and upload usage data to servers, allowing authorized caregivers or the patient to observe compliance records. This trial will evaluate MedSignals' usability and functionality in increasing medication compliance in people infected with HIV.

Participants will be randomly assigned to one of three study groups; each group will contain 25 participants. One group will use MedSignals with all of its features, one group will use MedSignals with only alarm features, and the final group will not use any device. Participants will have 4 study visits over 9 weeks and one follow-up telephone call after 6 months. Assessments will include demographic and usability questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected for at least six months prior to study entry
* Currently taking at least one and not more than four antiretroviral medications (not including medications for prophylaxis or unrelated disorders)
* Understand the benefits of antiviral medications in reducing viral load, boosting immune response, and preventing opportunistic infections
* Desire to take all antiretroviral medication as scheduled
* Working telephone
* Ambulatory
* Good mental health

Exclusion Criteria:

* Require assistance dispensing or taking medications
* Require full or part time assistance with the activities of daily living
* Does not intend to take all anti-HIV medication over the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2003-10; Primary Completion 2007-06 (Actual); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Medsignals performance | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Vesta Brue, MBA, Principal Investigator — Chairman
Locations (1):
- LIFETECHniques, Inc., Santa Barbara, California, United States